CLINICAL TRIAL: NCT06732219
Title: A Single-Arm Pilot Trial for Mitigating Relapse of Severe Problem Behavior
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Collaborators: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Principal Investigator, John Michael Falligant, Assistant Professor, Auburn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21HD112724 (NIH)
Record Dates: First submitted 2024-12-09; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Challenging Behavior
Keywords: neurodevelopmental disorders; autism; challenging behavior
MeSH Terms: conditions — Neurodevelopmental Disorders; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Enhanced Teaching Arm (Experimental): Participants in this arm will receive a behavioral intervention designed to reduce challenging behaviors and improve skill acquisition. The intervention includes functional communication training (FCT) to teach appropriate communication responses, the use of extinction-correlated stimuli to signal changes in reinforcement conditions, terminal probe schedule thinning to systematically reduce the frequency of reinforcement, competing stimuli to minimize engagement in challenging behaviors during reinforcement delays, and caregiver fading to promote skill generalization and maintenance across naturalistic environments. These strategies will be tailored to individual needs and administered within structured sessions.
  Interventions: Behavioral: Functional Communication Training; Behavioral: Extinction-Correlated Stimuli; Behavioral: Caregiver Fading; Behavioral: Structured-Probe Schedule Thinning; Behavioral: Multiple-Context Generalization Training

INTERVENTIONS:
Behavioral: Functional Communication Training — Functional Communication Training (FCT) focuses on teaching an appropriate functional communicative response (FCR) to access the reinforcer maintaining severe problem behavior (SPB). This procedure involves selecting an appropriate topography for the FCR (e.g., touching a card, exchanging a picture) and using a backward chaining approach. The training will progress from full physical prompts to partial prompts and eventually to independent, unprompted responses, all within a trial-based format.
Behavioral: Extinction-Correlated Stimuli — A distinct extinction-correlated stimulus (e.g., a laminated picture card) will be used in all treatment sessions where severe problem behavior (SPB) is subject to extinction contingencies. This stimulus will also be present during relapse challenges (described below). The selection of the stimulus will be individualized for each participant to ensure it has no prior association with treatment-related contexts, minimizing the influence of pre-existing learning histories.
Behavioral: Caregiver Fading — Behavioral Skills Training (BST) will be used to teach caregivers to (1) implement the behavioral intervention package (i.e., differential reinforcement of alternative behavior with extinction) in a controlled setting with confederates and (2) transition into behavioral sessions with the participant while gradually phasing out the clinical therapist.
  Caregivers will begin by implementing mastered intervention components alongside the therapist during sessions with the participant, where the therapist will provide in-situ feedback. Once the caregiver demonstrates at least 80% treatment integrity across two consecutive sessions, the therapist will systematically increase their distance by 3 meters each session (maintaining at least 80% integrity) until they are fully removed from the treatment area.
Behavioral: Structured-Probe Schedule Thinning — Once a clinically significant decrease in severe problem behavior (SPB) is achieved (defined as an 80% reduction from the baseline mean rate), schedule thinning will be implemented. This process involves reducing the density of reinforcement by introducing a multiple schedule with alternating periods where reinforcement for the functional communication response (FCR) is available and unavailable.
  Schedule thinning will begin immediately at the terminal schedule, with an 80% reduction in reinforcer density from treatment. Specifically, the FCR will be placed on extinction for 540 seconds and reinforced for 60 seconds during each session. This schedule was selected based on prior analyses of effective reductions in reinforcer density. If the treatment effect remains strong (defined as maintaining at least an 80% reduction in SPB relative to baseline), schedule thinning will proceed at this step until three consecutive sessions show consistent results.
Behavioral: Multiple-Context Generalization Training — In multiple-context training, treatment will be implemented at the terminal schedule (i.e., after completing schedule thinning) in new contexts, including unique locations and with different individuals, distinct from the setting used during the initial treatment phase.

SUMMARY:
The goal of this study is to improve how we teach self-control and communication skills to children and adolescents with challenging behaviors. Researchers aim to find ways to make behavior-change treatments more effective and long-lasting, even when the environment or reinforcement schedules change.

The main questions this study will answer are:

Can innovative techniques help children maintain learned skills, such as asking for attention or waiting for rewards, when faced with new people, places, or situations? How do cognitive and behavioral factors, like memory, timing, and decision-making, affect the success of treatments?

Participants in this study will:

Complete assessments to identify preferred activities and understand the causes of challenging behaviors.

Learn communication skills to replace challenging behaviors, such as tantrums or crying, with more appropriate actions like asking for attention.

Participate in activities designed to understand their individual responses to different types of rewards and delays.

DETAILED DESCRIPTION:
Purpose:

The purpose of this research is to explore experimental approaches for improving the durability and generalization of reinforcement-based behavioral interventions. While such interventions are highly effective for reducing challenging behaviors and teaching new skills, their effectiveness can diminish over time due to environmental changes, implementation inconsistencies, or reductions in reinforcement schedules. This study investigates how cognitive and behavioral factors influence treatment outcomes and tests innovative strategies to enhance the long-term success of behavior-change interventions.

Study Objectives:

Evaluate the feasibility of using innovative reinforcement-based tactics to enhance the durability of behavioral interventions.

Investigate how individual factors, such as timing perception, reward sensitivity, and decision-making, impact treatment outcomes.

Assess generalization and maintenance of newly acquired skills across various environmental contexts and with different individuals.

Methods and Procedures:

Participants will engage in a series of assessments and training sessions designed to identify and target challenging behaviors, replace them with functional communication skills, and evaluate the robustness of behavior change under varying conditions. The procedures include:

Preference Assessment:

Identifying preferred items and activities to use as reinforcers during treatment.

Competing Stimulus Assessment:

Identifying activities that engage participants during periods when high-preference items are unavailable.

Functional Behavioral Assessment:

Using interviews, direct observations, and experimental analyses to identify antecedents and consequences maintaining challenging behaviors, such as tantrums or crying.

Functional Communication Training (FCT):

Teaching participants alternative communication skills, such as requesting attention, that serve the same function as challenging behaviors.

Generalization and Maintenance Training:

Testing participants' ability to transfer learned skills to novel environments and individuals by systematically varying environmental contexts and reinforcement conditions.

ELIGIBILITY:
We will include individuals between the ages of 6 to 17 with IDD who have at least one topography of SPB that is maintained by social positive (e.g., attention, access to preferred items) reinforcement. The age range is driven by the need to maximize the number of participants; there is no evidence to suggest that age is a relevant variable regarding relapse of SPB.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Renewal and Resurgence of Challenging Behavior | From enrollment to the end of the intervention at 16 weeks
  The prevalence and magnitude of relapse (e.g., renewal or resurgence) in severe problem behavior (SPB). To assess relapse, we will calculate the highest single-session rate of SPB from the five most recent treatment sessions before a context change or reinforcement downshift (prechange period) and up to the first three sessions after the change (postchange period). If fewer sessions are available in either period, all available data will be used. Relapse will be identified if the maximum rate of SPB in any postchange session exceeds the maximum rate observed during all prechange sessions. The magnitude of relapse will be quantified using the log proportion rate of response, which normalizes session-by-session rates and allows for proportional comparisons across individuals. Outcome data will be collected during schedule thinning, generalization, and treatment challenges and compared to pooled relapse data from external controls to provide a benchmark for interpretation

CONTACTS AND LOCATIONS:
Overall Officials: John Falligant, PhD, Principal Investigator — Auburn University
Locations (2):
- United States (2):
  - Auburn University, Auburn, Alabama
  - Kennedy Krieger Institute, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Strohmeier CW, Cengher M, Chin MD, Falligant JM. Application of a terminal schedule probe method to inform schedule thinning with multiple schedules. J Appl Behav Anal. 2024 Jul;57(3):676-694. doi: 10.1002/jaba.1081. Epub 2024 May 9. PMID 38724468